CLINICAL TRIAL: NCT01925430
Title: The Evaluation of a New Sleep/Wake State Algorithm
Brief Title: The Evaluation of a New Sleep Algorithm
Status: Completed | Type: Observational
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Other Study IDs: MA06082013
Record Dates: First submitted 2013-08-15; First posted 2013-08-19 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2014-05

CONDITIONS: Healthy
Keywords: Observational; Sleep; Algorithm
MeSH Terms: interventions — Actigraphy

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Comparative product: A device which monitors sleep/wake states
  Interventions: Device: Comparative product
- Screening device: This device will screen for sleep-breathing disorders
  Interventions: Device: Screening device

INTERVENTIONS:
Device: Screening device — Non-invasive device worn over clothes during sleep. Used to screen for sleep-disordered breathing conditions.
  Other Names: ApneaLink; Actigraphy
  Groups: Screening device
Device: Comparative product — A non-invasive device worn on the arm or leg. It monitors body movement and sleep/wake states
  Other Names: Actiwatch 2 (Respironics); Patient data recorder; Actigraphy
  Groups: Comparative product

SUMMARY:
A new device is being developed to screen for sleep-breathing disorders. Within this device is a new software algorithm which will determine sleep/wake states. The aim of this study is to evaluate the performance of this new algorithm. This prototype will be compared against a commercially available device which monitors sleep/wake patterns. Volunteers will be asked to wear the prototype and comparative devices for 1-2 nights. The data from both devices will be downloaded after the completion of the study and analysis wil be performed to compare the two recordings.

ELIGIBILITY:
Inclusion Criteria:

* => 18yrs old
* can read and write English
* Provide informed written consent

Exclusion Criteria:

* Unable to participate for the full duration of the study
* An individual who is deemed unsuitable to participate in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteers who are employees within a medical device company
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2013-11; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Total sleep time | 12 hrs
  To measure the total sleep time recorded and analysed on the device using the new algorithm

SECONDARY OUTCOMES:
Frequency of arousals during sleep | 12 hrs
  To compare the data acquired of the new device's algorithm against a pre-existing device detailing the frequency of sleep and wake periods
Duration of arousals during sleep | 12 hrs
  To compare the data acquired of the new device's algorithm against a pre-existing device detailing the duration of sleep and wake
Occurrence of arousals during sleep | 12 hrs
  To compare the data acquired of the new device's algorithm against a pre-existing device detailing when sleep and wake periods occurred

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Schindhelm, BE PhD, Principal Investigator — The University of New South Wales, Australia & ResMed Ltd
Locations (1):
- RedMed Ltd, Sydney, New South Wales, Australia